CLINICAL TRIAL: NCT00373178
Title: Metabolic Effects of Treatment in Patients With Recently Diagnosed Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: University of Athens (Other)
Responsible Party: Principal Investigator, Nikolaos Kadoglou, MD,PhD, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 020401975
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: rosiglitazone; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone; Metformin

ARMS (1):
- Metformin,lifestyle counselling (Active Comparator)
  Interventions: Drug: rosiglitazone; Drug: metformin; Drug: Anti-diabetic medications

INTERVENTIONS:
Drug: rosiglitazone
Drug: metformin
Drug: Anti-diabetic medications

SUMMARY:
The aim of the present study is to investigate the influence of several anti-diabetic regimens (metformin,glitazone,sulfonylurea,glinidine) and diet on metabolic parameters in patients with recently diagnosed type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed type 2 diabetes
* No previous anti-diabetic medications

Exclusion Criteria:

* Heart failure
* Renal disease
* Liver disease
* Life-threatening diseases

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-01; Primary Completion 2007-01 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Novel cardiovascular risk factors modification | 2 years

SECONDARY OUTCOMES:
Lipid and glucose regulation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Miltiadis Alevizos, PhD, Study Chair — University Hospital AHEPA,Thessaloniki,Greece
Locations (2):
- Greece (2):
  - AHEPA University Hospital of Thessaloniki, Thessaloniki
  - Aristotle University of Thessaloniki, Thessaloniki

REFERENCES:
- [Derived] Gnesin F, Thuesen ACB, Kahler LKA, Madsbad S, Hemmingsen B. Metformin monotherapy for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Jun 5;6(6):CD012906. doi: 10.1002/14651858.CD012906.pub2. PMID 32501595
- [Derived] Kadoglou NP, Tsanikidis H, Kapelouzou A, Vrabas I, Vitta I, Karayannacos PE, Liapis CD, Sailer N. Effects of rosiglitazone and metformin treatment on apelin, visfatin, and ghrelin levels in patients with type 2 diabetes mellitus. Metabolism. 2010 Mar;59(3):373-9. doi: 10.1016/j.metabol.2009.08.005. Epub 2009 Oct 7. PMID 19815243